CLINICAL TRIAL: NCT00879645
Title: A Phase I Study to Assess the Pharmacokinetics of IK-1001 (Sodium Sulfide) in Subjects With Impaired Renal Function Following a Continuous 3-hour Intravenous Infusion
Brief Title: Pharmacokinetic Assessment of Sodium Sulfide in Subjects With Impaired Renal Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to develop a rapid & reliable assay to detect sulfide concentrations
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S103
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-10

CONDITIONS: Renal Impairment
Keywords: Renal Impairment; Renal Disease; Sodium Sulfide
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — sodium sulfide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sodium Sulfide - Mild Cohort (Experimental): Mild renal impairment (RI) Cohort administered 1.5 mg/kg/hr infusion of Sodium sulfide intravenously for 3 hours.
  Interventions: Drug: Sodium Sulfide
- Sodium Sulfide - Healthy Cohort (Experimental): Healthy subjects received sodium sulfide intravenously at 1.5 mg/kg/hr for 3 hours
  Interventions: Drug: Sodium Sulfide
- Sodium Sulfide - Moderate Cohort (Experimental): Moderate RI cohort received sodium sulfide intravenously at 1.5 mg/kg/hr for 3 hours
  Interventions: Drug: Sodium Sulfide
- Sodium Sulfide - Severe Cohort (Experimental): Severe RI cohort received sodium sulfide intravenously at 1.0 mg/kg/hr for 3 hours
  Interventions: Drug: Sodium Sulfide

INTERVENTIONS:
Drug: Sodium Sulfide — Sodium sulfide administered intravenously at 1.5 mg/kg/hr for 3 hours
  Other Names: IK-1001
  Arms: Sodium Sulfide - Mild Cohort
Drug: Sodium Sulfide — Sodium sulfide intravenously at 1.5 mg/kg/hr for 3 hours
  Other Names: IK-1001
  Arms: Sodium Sulfide - Healthy Cohort
Drug: Sodium Sulfide — Sodium sulfide intravenously at 1.5 mg/kg/hr for 3 hours
  Other Names: IK-1001
  Arms: Sodium Sulfide - Moderate Cohort
Drug: Sodium Sulfide — Sodium sulfide intravenously at 1.0 mg/kg/hr for 3 hours
  Other Names: IK-1001
  Arms: Sodium Sulfide - Severe Cohort

SUMMARY:
This is a Phase 1 study to assess the pharmacokinetics (PK) of IK-1001 (sodium sulfide) in healthy volunteers as well as in subjects with varying degrees of impaired renal function. A total of 28 subjects will be enrolled into the study over a 6 month period. There will be 4 cohorts. The first cohort will consist of subjects with mild renal impairment, the fourth cohort will be subjects with intermediate renal impairment and the third cohort will be subjects with severe renal impairment and the second cohort will consist of normal healthy subjects. All subjects will receive the study drug for 3 hours as a single intravenous (IV) infusion and will be followed over a 7 day period.

DETAILED DESCRIPTION:
This is a Phase 1 pharmacokinetic study to assess the pharmacokinetics of IK-1001 in healthy volunteers as well as subjects with varying degrees of impaired renal function following a single intravenous infusion.

A total of 28 subjects will be enrolled into the study, including 6 normal subjects (Creatinine Clearance (CrCL) > 80 mL/min), 9 subjects with mild impairment (CrCL ≥ 50 to < 80 mL/min), 6 subjects with intermediate impairment (≥ 30 to < 50 mL/min) and 7 subjects with severe impairment (CrCL < 30 mL/min).

Mild, moderate and normal healthy subjects will receive IK-1001 as a single IV infusion for 3 hours at 1.5 mg/kg/hr. Blood, plasma, urine and exhaled air will be collected from each subject over 48 hours and at follow-up visit (Day 7), to evaluate pharmacokinetics of Hydrogen Sulfide (H2S) (exhaled air), IK-1001 (blood) and thiosulfate in plasma and urine. Severe subjects will receive IK-1001 as a single IV infusion for 3 hours at 1.0 mg/kg/hr.

For each dosing cohort, the study will consist of a screening visit (Days -28 to -1), a treatment visit (Day 0 (check-in) to Day 3), and a follow-up (exit) visit day 7 (+/- 2 days).

Study subjects will be enrolled to one of 4 cohorts and all will receive investigational product at the given dose level. The subjects will be considered to be enrolled in the study at randomization.

IK-1001 will be administered by a healthcare professional intravenously over 3 hours using an infusion pump. Dosage of IK-1001 will be administered on actual body weight basis, according to cohort assignment and using the subject's body weight determined on Day -1. After the end of the initial 3-hour study period, subjects will be observed for an additional 45 hour period before discharge from the unit.

ELIGIBILITY:
Inclusion Criteria:

1. For normal subjects arm (CrCL > 80 ml/min): Healthy male and female subjects age 18 to 70 years of age inclusive. Pregnant women are excluded and women of child-bearing potential must agree to the use of medically reliable contraceptive methods for the duration of the study and for 30 days after study.

   For renally impaired arm: Male and female - pregnant women are excluded and women of child-bearing potential must agree to the use of medically reliable contraceptive methods for the duration of the study and for 30 days after study. Subjects with mild, moderate and severe renal function aged between 18 to 70 years old
2. Body mass index (BMI) within the range of 18 to 40 kg/m2
3. Electrocardiogram (ECG) recording without clinically relevant abnormalities
4. Having had no febrile or infectious disease for at least seven days prior to dosing of study drug
5. Able to communicate well with the study staff and to understand and comply with the requirements of the study, understand and sign the written informed consent

Exclusion Criteria:

1. High risk patients who may need an urgent dialysis during clinical conduct portion of the study (from Day -1 until last PK sampling on Day 7)
2. All smokers.
3. More than moderate alcohol consumption (>35 g ethanol regularly or > 2 drinks per day )
4. Any history of alcohol or drug abuse
5. Any active physical or psychiatric disease, acute or chronic
6. Any clinically relevant history of drug hypersensitivity, asthma, urticaria or other severe allergic diathesis
7. Pregnant or nursing women
8. Blood donation within 30 days
9. Participation in any clinical study within 30 days prior to the treatment phase of this study
10. Lab values outside of reference range and clinically relevant liver function tests (AST, ALT, gamma-GT)
11. Positive tests for HIV antibodies, Hepatitis B-virus surface antigen (HBsAg), Anti-Hepatitis C-virus antibodies (Anti-HCV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brahm Goldstein, MD, Study Director — Mallinckrodt
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Sulfide - Healthy Cohort: Healthy subjects received soduim sufide intravenously at 1.5 mg/kg/hr for 3 hours
Period: Overall Study
Arm/Group | Sodium Sulfide - Mild Cohort | Sodium Sulfide - Healthy Cohort | Sodium Sulfide - Moderate Cohort | Sodium Sulfide - Severe Cohort
Started | 9 | 6 | 6 | 7
Completed | 8 | 6 | 6 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Sulfide - Mild Cohort | Sodium Sulfide - Healthy Cohort | Sodium Sulfide - Moderate Cohort | Sodium Sulfide - Severe Cohort | Total
Number analyzed (Participants) | 9 | 6 | 6 | 7 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 6 | 7 | 28
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (7.41) | 56.1 (14.69) | 60.6 (7.91) | 48.9 (11.96) | 55.3 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 5 | 14
  Male | 6 | 3 | 3 | 2 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 6 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Thiosulfate in Plasma
Description: Total concentration of thiosulfate in plasma was measured through pharmacokinetic blood sampling.
Time Frame: 8 hours after treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Sulfide - Mild Cohort | Sodium Sulfide - Healthy Cohort | Sodium Sulfide - Moderate Cohort | Sodium Sulfide - Severe Cohort
Number analyzed (Participants) | 9 | 6 | 6 | 7
ng/mL | 120.4 (57.83) | 199.6 (100.74) | 199.1 (60.32) | 190.1 (36.41)

2. Primary Outcome: Thiosulfate in Urine
Description: Total concentration of thiosulfate in urine was measure through pharmacokinetic urine collection
Time Frame: 48 hours after treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Sulfide - Mild Cohort | Sodium Sulfide - Healthy Cohort | Sodium Sulfide - Moderate Cohort | Sodium Sulfide - Severe Cohort
Number analyzed (Participants) | 9 | 6 | 6 | 7
ng/mL | 1805.5 (552.00) | 2137.7 (688.83) | 1114.3 (720.79) | 603.8 (433.44)

3. Primary Outcome: Sodium Sulfide in Blood
Description: Total concentration of sodium sulfide in blood was measured through pharmacokinetic blood sampling.
Time Frame: 8 hours after treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Sulfide - Mild Cohort | Sodium Sulfide - Healthy Cohort | Sodium Sulfide - Moderate Cohort | Sodium Sulfide - Severe Cohort
Number analyzed (Participants) | 9 | 6 | 6 | 7
ng/mL | 51.2 (12.23) | 49.6 (14.58) | 49.8 (17.23) | 42.9 (5.55)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 6-month duration of the trial.
Description: Clinically significant changes in vital signs and laboratory values are recorded as adverse events.
Arm/Group | Sodium Sulfide - Mild Cohort | Sodium Sulfide - Healthy Cohort | Sodium Sulfide - Moderate Cohort | Sodium Sulfide - Severe Cohort
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 7/9 | 1/6 | 5/6 | 4/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Sulfide - Mild Cohort (N=9) | Sodium Sulfide - Healthy Cohort (N=6) | Sodium Sulfide - Moderate Cohort (N=6) | Sodium Sulfide - Severe Cohort (N=7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Paraesthesia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Phlebitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Site Anaesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application Site Irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application Site Rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Site Irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other